CLINICAL TRIAL: NCT05295212
Title: A Prospective, Multicenter Phase II Clinical Study of Atezolizumab Combined With Platinum-based Chemotherapy as Neoadjuvant Therapy for Patients With Resectable Stage II-IIIB Driver Gene-negative Non-small Cell Lung Cancer (NSCLC)
Brief Title: Atezolizumab Combined With Platinum-based Chemotherapy as Neoadjuvant Therapy for Patients With Resectable Stage II-IIIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NATAL
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (No Intervention): MRD revealed negative
- Cohort B (Experimental): MRD revealed positive
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Pemetrexed (500mg/m2)/Paclitaxel (260mg/m2) Carboplatin (AUC=4-5) Atezolizumab(1200mg) ivgtt, every 21 days Range from 4 cycles
  Arms: Cohort B

SUMMARY:
This study aimed to evaluate the efficacy, safety, tolerability, feasibility of surgery, and incidence of preoperative and postoperative complications of atezolizumab in combination with platinum-based chemotherapy with resectable stage II-IIIB non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects selected for this study must meet all of the following criteria:

  1. Sign written informed consent before implementing any trial-related procedures;
  2. Age ≥18 years old and ≤75 years old; No limit on the gender;
  3. Previously untreated, histologically confirmed resectable stage II, IIIA, IIIB (N2) (AJCC stage VIII) NSCLC; cTNM stage can be confirmed by PET-CT or pathological biopsy; resectable stage II non-small cell lung cancer is defined as radical resection as assessed by a qualified thoracic surgeon; resectable is resectable and potentially resectable as defined by the Expert Consensus on Multidisciplinary Diagnosis and Treatment of Stage III Non-small Cell Lung Cancer (2019 version); resectable includes IIIA (N0-1), some single-station mediastinal lymph node metastases with N2 and some T4 (satellite nodules present in adjacent lobes) N1; potentially resectable includes some stage IIIA and IIIB, including single-station N2 mediastinal lymph node short diameter < 3 cm stage IIIA NSCLC, potentially resectable T3 or T4 central tumors; Solid/solid pulmonary nodules, not pure ground-glass opacity (GGO), are strongly recommended for pathological puncture verification;
  4. Patients diagnosed with squamous cell carcinoma do not require genetic testing, and if they test positive for EGFR, ALK or ROS1, they are considered as exclusion criteria; if they are adenocarcinoma, they must undergo genetic testing containing at least EGFR, ALK and ROS1, and the acceptable detection method is ARMS or NGS, of which NGS is a cFDA-approved kit;
  5. Measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1;
  6. Twenty tissue sections (4-6 microns in thickness) should be submitted before enrollment for biomarker evaluation (tumor tissue samples must be fresh or archival samples obtained within 3 months before enrollment; fresh tissues must be biopsy specimens by hollow needle aspiration, resection or incision);
  7. ECOG score 0-1;
  8. Good organ function: (1) hematology: absolute neutrophil count (ANC) ≥ 1500/μL; platelets ≥ 100,000/μL; hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L; (2) kidney: serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cock-Gault formula); (3) liver: total bilirubin ≤ 1.5 × ULN or for subjects with total bilirubin levels > 1.5 × ULN, direct bilirubin is within normal limits; AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN; (4) endocrine system: thyroid stimulating hormone (TSH) is within normal limits. Note: If TSH is not within normal range at baseline, if T3 and free T4 are within normal range, then the subject can still meet the inclusion criteria; (5) Coagulation function: international normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, except: subjects receiving anticoagulant therapy, as long as PT or aPTT is within the proposed use range of anticoagulant drugs; (6) Cardiac function tests: baseline ECG showed no PR interval prolongation or atrioventricular block;
  9. The total lung function can withstand the proposed pneumonectomy surgery according to the surgeon's assessment;
  10. Women should agree to use contraceptive measures (such as intrauterine device (IUD), contraceptives or condoms) during the study and within 6 months after the end of the study; serum or urine pregnancy test is negative within 7 days before study entry, and must be non-lactating patients; men should agree to use contraceptive measures during the study and within 6 months after the end of the study period.

Exclusion Criteria:

* Subjects who meet the following criteria cannot be selected for this study:

  1. Histopathology is neuroendocrine carcinoma and sarcomatoid tumor；
  2. The presence of locally advanced unresectable or metastatic disease; unresectable including stage III non-small cell lung cancer multidisciplinary diagnosis and treatment expert consensus (2019 version) defined unresectable, including partial IIIA, IIIB and all IIIC, usually including single-station N2 mediastinal lymph nodes short diameter ≥ 3 cm or multi-station lymph nodes fused into a mass (CT lymph nodes short diameter ≥ 2 cm) N2, invading the esophagus, heart, aorta, pulmonary veins T4 and all N3;
  3. Subjects with known EGFR mutations or ALK, ROS1 translocations, non-squamous cell carcinoma subjects need to clarify the EGFR, ALK and ROS1 mutation status；
  4. Early stage NSCLC previously treated with systemic anticancer therapy, including treatment with investigational agents；
  5. History of (non-infectious) pneumonia/interstitial lung disease requiring steroid therapy, or current pneumonia/interstitial lung disease requiring steroid therapy；
  6. Known history of active tuberculosis;
  7. Known active infection requiring systemic treatment;
  8. Any known or suspected autoimmune disease or immunodeficiency subjects, except: patients with a history of hypothyroidism, if hormone therapy is not required, or are receiving physiological doses of hormone replacement therapy; subjects with stable type I diabetes whose blood glucose is controlled;
  9. Subjects with active hepatitis B (defined as positive hepatitis B virus surface antigen [HBsAg] test results and HBV-DNA test values higher than the upper limit of normal of the laboratory of the study site) or hepatitis C (defined as positive hepatitis C virus surface antibody [HCsAb] test results and positive HCV-RNA test results during the screening period);
  10. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive);
  11. Live vaccines within 30 days prior to the first dose. Including but not limited to the following: mumps, rubella, measles, varicella/herpes zoster (chickenpox), yellow fever, rabies, bacillus Calmette-Guerin (BCG) and typhoid vaccines (inactivated viral vaccines are allowed);
  12. Have ≥ grade 2 peripheral neuropathy;
  13. Previous treatment with PD-1/PD-L1 drugs or treatment with another drug targeting T cell receptor (such as CTLA-4, OX-40, etc.);
  14. Patients with any severe and/or uncontrolled diseases, such as: (1) unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmia; patients with unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); (2) active or uncontrolled severe infection; (3) liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis; (4) poor control of diabetes (fasting blood glucose (FBG) > 10 mmol/L); (5) urine routine showed urine protein ≥ + +, and confirmed 24-hour urine protein > 1.0g; (6) a history of psychiatric drug abuse and can not quit or mental disorders;
  15. Use of immunosuppressive drugs 2 times before the first study drug treatment, excluding topical glucocorticoids or systemic glucocorticoids no more than 10 mg/day prednisone or equivalent doses of other glucocorticoids;
  16. Pregnant or lactating women;
  17. Prisoners who are unlawfully incarcerated or compulsorily detained for non-mental illness or physical (such as infectious diseases) diseases;
  18. Patients with bleeding tendency (such as active gastrointestinal ulcers) or treatment with anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues;
  19. History of allergy to study drug ingredients;
  20. According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MPR Rate | 1.5 year
  Major pathological remissions
MRD negative Rate | 1.5 year
  Minimal residual disease rate

SECONDARY OUTCOMES:
pCR | 1.5 year
  Defined as the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) to the total subjects
DFS | 1.5 year
  disease-free survival
EFS | 1.5 year
  event-free survival
ORR | 1.5 year
  Overal response rat
OS | 1.5 year
  Overall survival time

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China